CLINICAL TRIAL: NCT00306904
Title: A Phase II, Pharmacokinetic, Randomized, Double-Masked, Controlled, Dose Comparison Study of Cand5 for Intravitreal Injection for the Treatment of Diabetic Macular Edema
Brief Title: Safety and Efficacy Study of Small Interfering RNA Molecule (Cand5) to Treat Diabetic Macular Edema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OPKO Health, Inc. (Industry)
Responsible Party: Denis O'Shaughnessy, Opko Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACU211
Record Dates: First submitted 2006-03-23; First posted 2006-03-27 (Estimated); Last update posted 2008-07-25 (Estimated); Status verified 2008-07

CONDITIONS: Diabetic Macular Edema
Keywords: Macular; Edema; Diabetic; Retinopathy
MeSH Terms: conditions — Edema; Retinal Diseases | interventions — bevasiranib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): 3.0 mg/eye dose group
  Interventions: Drug: bevasiranib
- 2 (Experimental): 1.5 mg/eye dose group
  Interventions: Drug: bevasiranib
- 3 (Experimental): 0.2 mg/eye dose group
  Interventions: Drug: bevasiranib

INTERVENTIONS:
Drug: bevasiranib
  Other Names: Cand5

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics, safety and preliminary efficacy of 3 doses of Cand5. Cand5 is a small interfering RNA molecule that selectively silences the mRNA encoding for VEGF. The target population are patients with diabetic macular edema.

DETAILED DESCRIPTION:
Diabetic retinopathy is the leading cause of newly diagnosed blindness in the working age (20-74) population in the United States1 and diabetic macular edema (DME) is the leading cause of vision loss in diabetic retinopathy. DME is the result of the breakdown of the retinal capillary endothelium in patients with diabetes mellitus (Type I and II).

A key factor in the development of DME is the permeability of the blood-retinal barrier. The breakdown of the endothelial tight junctions of the capillary walls in the retinal vasculature leads to increased permeation of salts, proteins, and water from the capillary luminal side of the barrier and the accumulation of fluid in the extracellular space. Multiple agents appear to contribute to the disruption of the blood-retina barrier,including vasoactive agents, prostaglandin and vascular endothelial growth factor (VEGF). VEGF is a peptide that promotes neovascularization and increases vascular permeability. If the resulting fluid is more than the amount that can be removed through the active pump mechanism (retinal pigmented epithelium), fluids continue to accumulate and edema develops. When thickening evolves or threatens the center of the fovea there is a high risk of visual loss.

Cand5 is a synthetic double stranded RNA (dsRNA) oligonucleotide. The molecule is a duplex formed by the hybridization of two partially complementary single strand RNAs in which the 3' end are capped with 2 deoxyribose (dT) units. Hybridization occurs across 19 ribose base pairs to yield the Cand5 molecule. Cand5 has a molecular weight of 13,345 grams/mole. Cand5 selectively silences the mRNA encoding for VEGF.

A comparison will be made between the three (3) treatment arms with regard to safety, efficacy, and duration of effect to determine a safe and efficacious dose of Cand5 appropriate for evaluation in future pivotal trials.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be male or female age 21 or older.
2. Patient must sign (and be given) a copy of the written informed consent form.
3. Patients must have the diagnosis of diabetes mellitus (type 1 or type 2). Patients with the following will be considered to be sufficient evidence that diabetes is present:

   * Current regular use of insulin for the treatment of diabetes mellitus OR
   * Current regular use of oral anti-hyperglycemia agents for the treatment of diabetes OR
   * Documented diabetes by WHO criteria
4. Patients must have ETDRS best corrected visual acuity of 69 to 24 letters (20/40 to 20/320 Snellen Equivalent) in the study eye.
5. Patients must have a mean retinal thickness on OCT ≥ 250 microns in the central subfield.

Exclusion Criteria:

1. Patients with a history of chronic renal failure requiring dialysis or kidney transplant.
2. A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure and glycemic control), including:

   * Patients in poor glycemic control who, within the last 4 months, initiated intensive insulin treatment (a pump or multiple daily injections) or plan to do so in the next 4 months should not be enrolled.
   * Patients with HbA1C > 10%OR
   * Patients with systolic blood pressure greater than 170 mmHg and/or diastolic blood pressure greater than 100 mmHg (Note: If blood pressure is brought below 170/100 mmHg by anti-hypertensive treatment, patient can become eligible).
3. Past panretinal photocoagulation (PRP) for diabetes within 12 weeks of screening or PRP expected to be needed in the next three months in the study eye.
4. Focal laser therapy to the retina of the study eye within 12 weeks of screening.
5. Any intraocular surgery or ocular laser procedures in the study eye within 12 weeks of screening.
6. Participation in an investigational trial within 30 days of study entry that involved treatment with any drug that has not received regulatory approval at the time of study entry.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-01; Primary Completion 2007-09 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline at the 12-week evaluation in macular edema as measured by optical coherence tomography.

SECONDARY OUTCOMES:
Mean BCVA line/letters change from baseline at the 12-week evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Du Castel, MD, Study Director — Chiltern International
Locations (1):
- Retina Associates of Cleveland, Beechwood, Ohio, United States

REFERENCES:
- See also: Sponsor — http://www.opko.com